CLINICAL TRIAL: NCT06461780
Title: Exploring Physical and Psychological Distress, Financial Toxicity, Care Needs and Quality of Life in Patients Receiving Immunotherapy in One Year Follow-up
Brief Title: Exploring Physical and Psychological Needs and Quality of Life in Patients With Advanced Cancer Receiving Immunotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023-03-005BC
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Immunotherapy; IrAE; Distress, Emotional; Care Need; Financial Toxicity; Quality of Life
MeSH Terms: conditions — Neoplasms; Financial Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The Line-based questionnaire follow-up app will be used to collect and follow patients' condition and syndrome.
  Interventions: Other: Line-based questionnaire follow-up

INTERVENTIONS:
Other: Line-based questionnaire follow-up — The participant will use LINE group to report irAE severity, distress, financial toxicity and change trajectory of quality of life in one-year follow-up. If the severity grade of irAE reach the threshold and require referral, an alarm will appear to notify the research team to conduct and transfer to a clinical specialitst, or refer to the emergency room for treatment. Additionally, the Line group will also provide clinical relevant immunotherapy health education information currently and routinely used in study site. Patients can view it according to their interests, but the APP will not actively promote it.

SUMMARY:
During the immune checkpoint inhibitor therapy (ICIT), most of the patients stay at home, but there is lacking of the studies to explore their physical and psychological distress, financial toxicity, care needs, and quality of life. Therefore, the aims of this program are to (1) explore the immune-related adverse event (irAE) severity, distress, financial toxicity, and quality of life and examine the psychometric testing of the Functional Assessment of Cancer Therapy-Immune Checkpoint Modulator (FACT-ICM); (2) establish the LINE group for assessing irAE severity and change trajectory of quality of life in one-year follow-up and (3) combined retrospective chart review and the finding in aim (2) to develop the risk prediction model in order to identify the high risk population.

DETAILED DESCRIPTION:
To achieve aim 1, a cross-sectional design is conducted to explore irAE severity, distress, financial distress, and quality of life in mixed type of cancer patients receiving ICIT. A structural questionnaire will be used including Common Terminology Criteria for adverse events (CTCAE) 33 items, Distress Thermometer (DT), the Comprehensive Score for financial Toxicity (COST), FACT-ICM, and EORTC-QLQ C30. Correlation analysis and exploratory factor analysis will be used to examine the psychometric testing of FACT-ICM.

To achieve aim 2 and 3, a prospective cohort study will be conducted to recruit 200 patients in first course receiving ICIT and follow for 1 year using LINE to report symptoms in weekly reporting within 3 months and once in 3-4 weeks in 4th -12th months during treatment. Data will be collected at five times (Before treatment for baseline, the 3th, 6th 9th 12th months) using a set of questionnaires including CTCAE 33 items, DT, COST, Supportive Care Needs Scale-short form34, and FACT-ICM.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients diagnose cancer and are informed
* (2) Aged ≥18 years old
* (3) Conscious clear and able to communicate

Exclusion Criteria:

* (1) Patients who are under other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient-Report Outcome-- Common Terminology Criteria for adverse events (PRO-CTCAE) | The data will be collected once a week within 3 months and once in 3-4 weeks in 4th-12th months during treatment.
  Interviewers graded the severity of adverse events according to the Common Terminology Criteria for adverse events (CTCAE), version 5, from the National Cancer Institute (NCI). In this study, we included 33 important symptoms from PRO-CTCAE in immunotherapy patients.
Symptom Severity Scale (SSS) | The data will be collected at five times (Before treatment for baseline, the 3rd, 6th, 9th, and 12th month)
  The Symptom Severity Scale (SSS) was used to evaluate the symptom severity of cancer patients. It included 25 common symptoms in cancer patients.The severity was scored by an 11-point numerical rating scale, from 0 (not at all) to 10 (very severe).
Distress Thermometer (DT) | The data will be collected at five times (Before treatment for baseline, the 3rd, 6th, 9th, and 12th month)
  The Distress Theremometer is utilized to assess patients' emotional distress and its sources. The assessment was developed by National Comprehensive Cancer Network (NCCN) and to evaluate the psychological distress level of cancer patients. It a single-item-11-point scale, from 0 to 10 points, which ask patients about their overall distress level over the past week, with higher scores indicating higher levels of distress.
The COmprehensive Score for financial Toxicity-Functional Assessment of Chronic Illness Therapy (COST-FACIT) | The data will be collected at five times (Before treatment for baseline, the 3rd, 6th, 9th, and 12th month)
  The COST-FACIT developed by Souza, is used to assess patients' financial distress. It evaluates the financial situation of patients undergoing treatment for chronic diseases. The scale consists of 12 items rated on a 0 to 4 Likert-type scale, where 0 indicates "not at all important" and 4 indicates "very important." Lower scores indicate greater financial toxicity.
The Functional Assessment of Cancer Therapy-Immune Checkpoint Modulator (FACT-ICM) | The data will be collected at five times (Before treatment for baseline, the 3rd, 6th, 9th, and 12th month)
  The FACT-ICM is used to assess the quality of life in cancer patients undergoing immunotherapy. It comprises 25 symptom-related items specific to immune checkpoint modulation therapy and 27 items from the Functional Assessment of Cancer Therapy-General (FACT-G), totaling 52 items. Ratings are done on a 0 to 4 Likert-type scale, where 0 indicates no distress at all and 4 indicates extreme distress.
European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire 30 (EORTC-QLQ-C30) | The data will be collected at five times (Before treatment for baseline, the 3rd, 6th, 9th, and 12th month)
  To assess the convergent validity of the FACT-ICM, we employed this scale to analyze the correlation between two sets of quality of life data. It consists of 30 items assessing five major functional domains in cancer patients. Ratings for most items are done on a 1 to 4 Likert-type scale, where 1 indicates no presence and 4 indicates very severe presence of symptoms, with higher scores indicating poorer quality of life.
Supportive Care Needs Survey-Short Form 34 (SCNS-SF34) | The data will be collected at five times (Before treatment for baseline, the 3rd, 6th, 9th, and 12th month)
  The SCNS-SF34 comprises 34 items and utilizes a 1 to 5 Likert-type scoring system, where 1 indicates no need and 5 indicates the greatest need for assistance. Scores for each domain, based on the total scores of individual items, are standardized to a range of 0 to 100, with higher scores indicating greater unmet needs in that domain.

CONTACTS AND LOCATIONS:
Overall Officials: I-Wen Chang, PHD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Based on the Institutional Review Board of the study site, the patients does not agree to give their data to other study.